CLINICAL TRIAL: NCT01306851
Title: Multicenter, Randomized, Controlled, Single Blinded, Phase IV Study Comparing 2 Parallel Groups in the Evaluation of the Prevention of Anastomotic Leaks in GI High Risk Anastomosis, With or Without the Application of Fibrin Glue in the Anastomotic Line
Brief Title: Prevention of Anastomotic Leak in Gastrointestinal (GI) Anastomosis With the Application of Tisseal in the Anastomotic Line
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital General Universitario Gregorio Marañon (Other)
Responsible Party: Jesús Lago Oliver, Hospital General Universitario "Gregorio Marañón"
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PROTTISUCOL-001
Record Dates: First submitted 2011-03-01; First posted 2011-03-02 (Estimated); Last update posted 2011-03-02 (Estimated); Status verified 2007-05

CONDITIONS: Anastomotic Leak
Keywords: fibrin glue; anastomotic leak; gastrointestinal high risk anastomosis
MeSH Terms: conditions — Anastomotic Leak | interventions — Fibrin Tissue Adhesive

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- Fibrin glue (Active Comparator)
  Interventions: Drug: Fibrin glue

INTERVENTIONS:
Drug: Fibrin glue — In the intervention group, 5 or 10 ml of fibrin glue are applied in the anastomotic line.

SUMMARY:
The anastomotic leak is one of the most feared complications in abdominal surgery. Certain control methods have been described but the incidence of that complication remains high and is the first cause of mortality in operations where gut anastomosis are performed.

With the aim to prove that the use of fibrin glue in the gut anastomosis can improve gut cicatrization, the investigators started the recruitment of patients to that clinical trial in 2007 with the study hypothesis that patients with a gut anastomosis where fibrin glue was used, had less anastomotic leaks than that where the fibrin glue was not used.

The investigators have calculated the number of patients necessaries to have statistical significant differences in 200 patients with a rate anastomotic leak expected to be higher than 10%.

The study include all the patients that usually arrive to our surgery department and that are expected to have a high risk gut anastomosis: rectal anastomosis, GI anastomosis in the obese patient, small bowel anastomosis in the obstructed one and esophageal anastomosis.

The study is randomized, simple blind where the patient does not know if they are in the fibrin glue group or not, and prospectively analyzed. All the clinical and laboratory or radiographic finds relative to the occurrence of an anastomotic leak are recorded.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing GI surgery where a high risk anastomosis is preview to be done

Exclusion Criteria:

* Haemodynamic instability
* Advanced oncologic disease
* Proteins below 4 gr/ml

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2007-06; Primary Completion 2013-03 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
Occurence of anastomotic leak | 6 months
  The occurence of anastomotic leak in the 6 months after the surgery is the most important factor to determine if fibrin glue is helpful in the prevention of that complicacion.

SECONDARY OUTCOMES:
Evidence of infectious collections in the anastomotic area | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital General Universitario Gregorio Marañon, Madrid, Madrid, Spain

REFERENCES:
- [Derived] Lago Oliver J, Arjona Medina I, Martin Garcia-Almenta E, Martin Gil J, Sanz Sanchez M, Perez Diaz MD, Alonso Poza A, Turegano Fuentes F, Torres Garcia A. [Use of fibrin based biological adhesives in the prevention of anastomotic leaks in the high risk digestive tract: preliminary results of the multicentre, prospective, randomised, controlled, and simple blind phase IV clinical trial: Protissucol001]. Cir Esp. 2012 Dec;90(10):647-55. doi: 10.1016/j.ciresp.2012.05.007. Epub 2012 Jun 27. Spanish. PMID 22748849